CLINICAL TRIAL: NCT00720876
Title: A Phase II Study of Vorinostat (Suberoylanilide Hydroxamic Acid) Plus Rituximab in Indolent Non-Hodgkin's Lymphoma
Brief Title: Vorinostat and Rituximab in Treating Patients With Indolent Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07195; P30CA033572 (NIH); CDR0000600989 (Registry Identifier: PDQ); NCI-2010-00531 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-07-22; First posted 2008-07-23 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — Rituximab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat and Rituximab (Experimental): Vorinostat by mouth two times (2X) per day for two weeks followed by one week of rest. Rituximab intravenously once every three weeks .
  Interventions: Biological: rituximab; Drug: vorinostat

INTERVENTIONS:
Biological: rituximab — Rituximab will be administered at a dose of 375 mg/m2 on day 1 of every cycle, every 3 weeks.
Drug: vorinostat — 200 mg twice daily, orally for 14 days followed by a seven day break on a 21 day cycle.

SUMMARY:
RATIONALE: Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving vorinostat together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects of giving vorinostat together with rituximab and to see how well it works in treating patients with indolent non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the anti-tumor activity of vorinostat and rituximab, in terms of objective response rate, time to progression, and survival, in patients with indolent non-Hodgkin lymphoma.
* To assess the toxicity profile of this regimen in these patients.

OUTLINE: Patients receive oral vorinostat twice daily on days 1-14 and rituximab IV on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

Patients must have histologically or cytologically confirmed indolent Non-Hodgkin's Lymphoma; included in this category are newly diagnosed or relapsed/refractory follicular center lymphomas grade I, II, III, relapsed/refractory marginal zone B-cell lymphoma (nodal and extranodal), relapsed/refractory mantle cell lymphoma

Patients must have measurable disease by computed tomography (CT) scan; positron emission tomography (PET) scan evaluations are desirable but not mandatory, so that patients with negative PET scans but measurable disease by CT are eligible

Patients may have had up to four prior chemotherapeutic regimens; steroids alone and local radiation do not count as regimens (radiotherapy must have been completed at least 14 days prior to starting vorinostat); Rituxan alone does not count as a regimen; however, Bexxar or Zevalin do; for treated patients, the most recent therapy must have failed to induce a complete response (i.e., there is persistent disease by CT or PET), or there must be disease progression or recurrence after the most recent therapy

Patients may be enrolled who relapse after autologous stem cell transplant if they are at least three months after transplant, and after allogeneic transplant if they are at least six month post transplant; to be eligible after either type of transplant, patients should have no active related infections (i.e., fungal or viral); in the case of allogeneic transplant relapse, there should be no active acute graft versus host disease (GvHD) of any grade, and no chronic graft versus host disease other than mild skin, oral, or ocular GvHD not requiring systemic immunosuppression

Life expectancy of greater than 3 months

Eastern Cooperative Oncology Group (ECOG) performance status 2 (Karnofsky >= 60%)

Absolute neutrophil count >= 1,000/mcL

Platelets >= 100,000/mcL

Total bilirubin within normal institutional limits; patients with elevation of unconjugated bilirubin alone, as in Gilbert's disease, are eligible

Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal

Creatinine up to and including 2 mg/dl

Pre-menopausal women must have a negative serum pregnancy test prior to entry on this study; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

Patients who have had chemotherapy within 4 weeks, or radiotherapy within 2 weeks or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are excluded; this does not include use of steroids, which may continue until two days prior to enrollment; low dose chlorambucil should be stopped two weeks prior to beginning vorinostat; valproic acid should be stopped at least two weeks prior to enrollment; nitrosoureas and mitomycin should be stopped 6 weeks prior to enrollment

Patients may not be receiving any other investigational agents

Patients with known brain metastases are excluded from this clinical trial unless the metastases are controlled after therapy and have not been treated with steroids within the past two months

History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat

There must be no plans for the patient to receive concurrent hormonal, biological, or radiation therapy

Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Pregnant women are excluded from this study; breastfeeding should be discontinued if mother is treated with vorinostat

Human immunodeficiency virus (HIV)-positive patients receiving combination antiretroviral therapy are ineligible; in addition, HIV patients not receiving combination antiretroviral therapy are also ineligible

Patients with other active malignancies are ineligible for this study

Patients with preexisting or previous coagulation issues are not excluded from study as long as 1) previous pulmonary embolism or deep vein thrombosis have been adequately treated or 2) if they are actively receiving Coumadin or lovenox for anticoagulation; patients who are already on coumadin or lovenox do not need to take additional 40 mg subcutaneous injections daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07-23 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chen, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California

REFERENCES:
- [Derived] Chen R, Frankel P, Popplewell L, Siddiqi T, Ruel N, Rotter A, Thomas SH, Mott M, Nathwani N, Htut M, Nademanee A, Forman SJ, Kirschbaum M. A phase II study of vorinostat and rituximab for treatment of newly diagnosed and relapsed/refractory indolent non-Hodgkin lymphoma. Haematologica. 2015 Mar;100(3):357-62. doi: 10.3324/haematol.2014.117473. Epub 2015 Jan 16. PMID 25596263

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vorinostat and Rituximab
Started | 30
Completed | 28
Not Completed | 2
Not completed — found to be ineligible after starting tx | 2

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat and Rituximab: Vorinostat by mouth 2X per day for two weeks followed by one week of rest. Rituximab intravenously once every three weeks .
  rituximab: Rituximab will be administered at a dose of 375 mg/m2 on day 1 of every cycle, every 3 weeks.
  vorinostat: 200 mg twice daily, orally for 14 days followed by a seven day break on a 21 day cycle.
Arm/Group | Vorinostat and Rituximab
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete and Partial Response)
Description: Response was assessed according to the 2007 Cheson criteria using CT scans or PET: Complete Response (CR), Disappearance of all evidence of disease; Partial Response (PR), >=50% decrease in the Sum of the Product of Diameters (SPD) of up to 6 largest dominant masses and no increase in the size of other nodes; Overall Response (OR) = CR + PR.
Time Frame: After every 3 cycles, up to 1 year after the start of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Vorinostat and Rituximab
Number analyzed (Participants) | 28
percentage of participants | 46

2. Secondary Outcome: Progression-free Survival
Description: Progression\Relapse is defined using the 2007 Cheson criteria, as appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy; or at least a 50% increase for nadir in the SPD of any previously involved nodes; or at least a 50% increase in the longest diameter of any singe previously identified node more than 1 cm in its short axis. Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until disease progress\relapse, up to 1 year after the start of treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vorinostat and Rituximab
Number analyzed (Participants) | 28
Months | 29.2 [14.4 to 51]

3. Secondary Outcome: Number of Participants With Grade 3 and 4 Toxicities
Description: Grade 3 & 4 toxicities at least possible related to study drugs during any cycle of treatment. Toxicity graded according to Common Terminology Criteria for Adverse Events version 3.0.
Time Frame: 3 weeks after the stop of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vorinostat and Rituximab
Number analyzed (Participants) | 28
Participants
  Neutrophil count decreased | 3
  Platelet count decreased | 5
  Hemoglobin decreased | 1
  Lymphocyte count decreased | 7
  Hypotension | 2
  Chills | 1
  Fatigue | 9
  Dehydration | 3
  Diarrhea | 1
  Kidney infection | 1
  Pneumonia | 2
  Sepsis | 1
  Urinary tract infection | 1
  Localized edema | 1
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Blood glucose increased | 3
  Serum phosphate decreased | 3
  Serum potassium decreased | 2
  Muscle weakness | 1
  Syncope | 1
  Hypoxia | 1
  Pneumonitis | 1
  Thrombosis | 4
  Vascular access complication | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of seven years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Vorinostat and Rituximab
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat and Rituximab (N=30)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 4 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat and Rituximab (N=30)
Hemoglobin decreased (Blood and lymphatic system disorders) | 22 (152)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (8)
Cardiac disorder (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (5)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (2)
External ear pain (Ear and labyrinth disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 4 (6)
Eye disorder (Eye disorders) | 2 (8)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (13)
Abdominal pain (Gastrointestinal disorders) | 13 (48)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 16 (50)
Diarrhea (Gastrointestinal disorders) | 24 (304)
Dry mouth (Gastrointestinal disorders) | 11 (27)
Dyspepsia (Gastrointestinal disorders) | 8 (19)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 10 (14)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 22 (174)
Oral hemorrhage (Gastrointestinal disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 2 (12)
Stomach pain (Gastrointestinal disorders) | 2 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (33)
Chest pain (General disorders) | 8 (9)
Chills (General disorders) | 16 (67)
Edema limbs (General disorders) | 11 (26)
Facial pain (General disorders) | 2 (3)
Fatigue (General disorders) | 26 (279)
Fever (General disorders) | 14 (26)
Flu-like symptoms (General disorders) | 2 (2)
Injection site reaction (General disorders) | 4 (4)
Localized edema (General disorders) | 4 (14)
Pain (General disorders) | 6 (8)
Hypersensitivity (Immune system disorders) | 8 (10)
Eye infection (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Lip infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 5 (17)
Tooth infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 8 (9)
Urinary tract infection (Infections and infestations) | 6 (12)
Wound infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 10 (13)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 6 (13)
Alanine aminotransferase increased (Investigations) | 11 (20)
Alkaline phosphatase increased (Investigations) | 10 (37)
Aspartate aminotransferase increased (Investigations) | 18 (54)
Bilirubin increased (Investigations) | 1 (9)
Creatinine increased (Investigations) | 18 (128)
Leukocyte count decreased (Investigations) | 16 (143)
Lymphocyte count decreased (Investigations) | 11 (49)
Neutrophil count decreased (Investigations) | 15 (75)
Platelet count decreased (Investigations) | 20 (137)
Weight loss (Investigations) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 19 (71)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (8)
Blood glucose increased (Metabolism and nutrition disorders) | 15 (55)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (9)
Serum albumin decreased (Metabolism and nutrition disorders) | 15 (45)
Serum calcium decreased (Metabolism and nutrition disorders) | 16 (51)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (11)
Serum glucose decreased (Metabolism and nutrition disorders) | 16 (90)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 5 (10)
Serum phosphate decreased (Metabolism and nutrition disorders) | 9 (16)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (14)
Serum potassium increased (Metabolism and nutrition disorders) | 9 (22)
Serum sodium decreased (Metabolism and nutrition disorders) | 15 (63)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (4)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (17)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (17)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Joint pain (Musculoskeletal and connective tissue disorders) | 8 (17)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 12 (16)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (6)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (4)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (66)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 12 (41)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 14 (58)
Memory impairment (Nervous system disorders) | 4 (8)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (14)
Speech disorder (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 10 (47)
Tremor (Nervous system disorders) | 3 (9)
Agitation (Psychiatric disorders) | 3 (7)
Anxiety (Psychiatric disorders) | 5 (24)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 5 (8)
Insomnia (Psychiatric disorders) | 9 (28)
Psychosis (Psychiatric disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (5)
Protein urine positive (Renal and urinary disorders) | 1 (2)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (7)
Urogenital disorder (Renal and urinary disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 12 (23)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (106)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (59)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (64)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 7 (15)
Sweating (Skin and subcutaneous tissue disorders) | 9 (13)
Flushing (Vascular disorders) | 2 (2)
Hemorrhage (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 8 (25)
Hypotension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT00720876/Prot_SAP_000.pdf